CLINICAL TRIAL: NCT02435628
Title: Relationship Between Psychosocial Factors, Health Literacy, Quality of Life and Satisfaction With Medical Visits in Adults With Neurofibromatosis 1, Neurofibromatosis 2, and Schwannomatosis
Brief Title: Relationship Between Psychosocial Factors, Health Literacy, Quality of Life and Satisfaction With Medical Visits in Adults With NF
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Clinical Psychologist, Massachusetts General Hospital
Other Study IDs: 2014P002755
Record Dates: First submitted 2015-04-29; First posted 2015-05-06 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Neurofibromatosis
MeSH Terms: conditions — Neurofibromatoses | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Satisfaction Questionnaires: After enrollment, subjects will be given baseline measures to assess demographics, psychosocial factors, and health literacy. This assessment will occur online via Computerized Assessment Center. Participants will complete the PROMIS battery of measures assessing: depression, anxiety, anger, fatigue, pain behavior and interference, physical function, satisfaction with discretionary social activities, satisfaction with social roles, and health literacy. Participants will also complete the FFFHL scale.
  Upon completion of the baseline assessments, the participant will meet with their doctor at the NF clinic for a routine appointment. Post-treatment assessments will be administered immediately after completion of the medical visit. This assessment will evaluate the participant's satisfaction with the appointment in the NF clinic using the MISS and CAHPS surveys. This will be done online via REDCap.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — All subjects will complete baseline psychological assessments prior to their medical visit. Upon completion of their routine medical visit, subjects will complete a post-test assessment measuring their satisfaction with the visit.

SUMMARY:
This is a prospective study through the NF clinic at Massachusetts General Hospital that will examine the relationship between psychosocial factors, health literacy, and satisfaction with the medical visit in adults with NF1, NF2, and Schwannomatosis. A total of 89 participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Can read and speak English at or above the 6th grade level
3. Diagnosis of neurofibromatosis type 1, neurofibromatosis type 2, or schwannomatosis

Exclusion Criteria:

1. Severe active or untreated major mental illness that would interfere with study participation, to be determined at the discretion of the study investigator (e.g. untreated psychosis or suicidality)
2. Unable or unwilling to participate
3. Unable or unwilling to complete psychological assessments online via the REDCap or Assessment Center systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with neurofibromatosis 1, neurofibromatosis 2, or schwannomatosis
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) | Baseline (pre-medical visit)
  A battery of measures assessing: depression, anxiety, anger, fatigue, pain behavior and interference, physical function, satisfaction with discretionary social activities, satisfaction with social roles, and health literacy.
Functional, Communicative and Critical Health Literacy (FFFHL) scale | Baseline (pre-medical visit)
  Measures one's health literacy, the capacity of individuals to access, understand, and use health information to make informed and appropriate health-related decisions.
Medical Interview Satisfaction Scale (MISS) | Participants will be followed for the duration of their medical visit, an expected average of no more than 2 hours.
  Measures patient satisfaction with individual doctor-patient consultations.
Consumer Assessment of Healthcare Providers and Systems (CAHPS) survey | Participants will be followed for the duration of their medical visit, an expected average of no more than 2 hours.
  Asks patients to report on and evaluate their experiences with health care. This survey covers topics that are important to consumers and focus on aspects of quality that consumers are best qualified to assess, such as the communication skills of providers and ease of access to health care services.

OTHER OUTCOMES:
Age, Gender, Ethnicity, and Race of Patients with NF | Baseline (pre-medical visit)
  The questionnaire asks for the patient's age, gender, ethnicity, and race as part of the basic demographics.
Visual Analog Health Scale | Participants will be followed for the duration of their medical visit, an expected average of no more than 2 hours.
  Measures one's current health on a scale from 0 ("very poor") to 10 ("very good").
Learning Disabilities of Patients with NF | Participants will be followed for the duration of their medical visit, an expected average of no more than 2 hours.
  This question asks patients if they have ever been diagnosed with a learning disability.
First Time at NF Clinic | Participants will be followed for the duration of their medical visit, an expected average of no more than 2 hours.
  This question asks the patient if it's their first time at the MGH NF clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States